The Use of Clear Aligners with Movement Enhancement Techniques NCT02087163

January 9, 2019

## Study Summary

| Title | The Use of Clear Aligners with Movement Enhancement Techniques |
|---|---|
| Objectives | Evaluated whether movement enhancement techniques increased the rate and length of tooth movement, and length of total treatment time. |
| Purpose | The purpose of this study was to use clear aligners to measure tooth |
| | movement and length of treatment. |
| Relevant Scientific | Orthodontic tooth movement is the result of forces applied to the crown of a |
| Background | tooth and the biological remodeling of the soft and hard tissues. |
| | The Invisalign® System (Align Technology, San Jose, California, USA) |
| | accurately fabricates removable clear aligners to move teeth with relative |
| | precision to provide comprehensive orthodontic treatment. Some |
| | practitioners advise patients to change aligners at 1-2 week wear time |
| | intervals in order to reduce treatment time or for other orthodontic or dental |
| | reasons. Animal studies in mice and rats have suggested that low magnitude, |
| | high frequency mechanical stimuli increases the healing of bony lesions in |
| | non-weight bearing bones, enhances the adaptive remodeling of condylar |
| | cartilage as evidenced by the advent of endochondral bone replacing |
| | hypertrophic cartilage, and enhances the effect of mechanical and magnetic |
| | forces on tooth movement. |
| Design | This was a non-significant risk, multicenter, randomized prospective study |
| | conducted at three sites in North America. A total of 90 adult patients who |
| | were eligible for Invisalign® Full treatment per the standard Invisalign® |
| | Instructions for Use were recruited for the study. Subjects were randomly |
| | placed into either a 7 day or 14 day aligner wear schedule. |
| Primary Outcome | Tooth movement change was calculated. |
| | <ul> <li>Participants were followed for the duration of orthodontic treatment,<br/>an average of 78 weeks.</li> </ul> |
| Secondary Outcome | Length of treatment change was calculated as number of clear aligners used. |
| | Participants were followed for the duration of orthodontic treatment, Participants wer |
| | an average of 78 weeks. |
| Treatment | Clear aligners with movement enhancement techniques. |
| · | |

| Eligibility Criteria | Inclusion Criteria: |
|---|---|
| | A subject were considered eligible if <u>all</u> of following inclusion criteria were fulfilled: |
| | Males or females between the ages of 16-46 inclusive |
| | Required orthodontic treatment |
| | Had permanent dentition |
| | No craniofacial anomaly present |
| | No past and present signs and symptoms of periodontal disease |
| | <ul> <li>No significant medical history or medication that would adversely<br/>affect the development or structure of the teeth and jaws and any<br/>subsequent tooth movement</li> </ul> |
| | No previous orthodontic or orthopaedic relapse |
| | No history of trauma, bruxism or parafunction |
| | No skeletal jaw discrepancy |
| | Angle Class I or Class II molar and canine relationship |
| | Crowding of at least 4mm per arch |
| | No osteoporosis drugs |
| | Exclusion Criteria: |
| | A subject was considered ineligible if <u>any</u> one of the following exclusion criteria were fulfilled: |
| | Subjects who did not fulfill all inclusion criteria requirements |
| Sites | 3 participating doctors in the North America. |
| Sample Size | 90 subjects. |
| Length of Study | Approximately 4 years. |
| Statistical Analysis | Pretreatment records were analyzed to measure the exact amount of |
| Plan | crowding. A discriminate analysis was used to ensure that there was no |
| | significant difference between study groups in any parameters (crowding, overjet, overbite, crossbite, gender, age, race,) that may have impacted the |
| | analysis of the efficacy of the aligners and the aligners with movement enhancement techniques. |
| | A multivariate analysis was conducted to determine if time or treatment modality showed an effect. |

| | Rate of tooth movement, length of treatment, and length of total treatment time were analyzed between all study groups. |
|---|---|
| | A sample size of 90 was selected to determine if future studies should be conducted based on the outcome of this study. |
| Results | Subject Enrollment |
| | <ul> <li>Started: 90 <ul> <li>70 female</li> <li>20 male</li> </ul> </li> <li>Completed: 73 <ul> <li>Not completed: 17</li> </ul> </li> <li>All 73 completed subjects were included in the data analysis which was conducted by Align's own statisticians. Tooth movement change was</li> </ul> |
| | measured as a millimeters of change per aligner. Length of treatment change was measured as the number of weeks. No Adverse Events were reported. |